CLINICAL TRIAL: NCT06333444
Title: The Role of Mentalization, Emotional Regulation and Loneliness in College Students' Psychological Distress
Brief Title: Counselling Intervention for College Students Experienced Psychological Distress
Acronym: TRESPASS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Alda Troncone, Principal Investigator, University of Campania Luigi Vanvitelli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: n. 08, 09/03/2021
Record Dates: First submitted 2024-03-19; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: University Students; Psychological Intervention; Psychological Distress
Keywords: university students; university counselling service; mental health; academic motivation
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Four weekly psychological counselling intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychological intervention (Experimental): four weekly psychological counselling intervention
  Interventions: Behavioral: four weekly psychological counselling intervention

INTERVENTIONS:
Behavioral: four weekly psychological counselling intervention — four weekly psychological counselling intervention delivered by university students asking help to university counselling service in Southern Italy

SUMMARY:
The goal of this clinical trial is to evaluate mental health and academic motivation in university students asking help to university counselling service (UCS) in Southern Italy before anf after four weekly psychological sessions.

The main question it aims to answer are:

* is the psychological counselling intervention useful in improving psychological distress and academic motivation
* which psychological variables predict the intervention outcome

DETAILED DESCRIPTION:
The participants will be university students who completed psychological counselling intervention delivered by UCS (University of Campania, Italy). They will be asked to completed an internet-based survey, administered anonymously through Google Forms. The survey consist of two sections. The first section includes questions about sociodemographic characteristics (e.g., gender and age), enrollment year, type of university course attended, academic standing (i.e., whether all exams within the prescribed period had been passed), and previous or current contact with psychological or psychiatric mental health services (university or non-university). The second section comprises four scales that assessed the variables of interest.

To measure psychological distress and problems, the Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) will be used. Feelings of loneliness will be assessed using the University of California-Los Angeles Loneliness Scale version 3 (UCLA-LS3). Emotion regulation will be assessed using the Difficulty in Emotion Regulation Scale (DERS). Students intentions to continue or to drop out of the academic course will be measured with self-reported questions.

ELIGIBILITY:
Inclusion Criteria:

* being university students who asked psychological help to university counselling service and completed the intervention

Exclusion Criteria:

* do not speak Italian

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
psychological distress | before and after the treatment, up to 7 weeks
  To measure psychological distress and problems, the Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) (Barkham et al., 1998; Evans et al., 2000). The CORE-OM is a 34-item self-report measure that evaluates the level of psychological distress will be used. The measure covers four domains: subjective well-being (4 items), problems/symptoms (depression: 4 items, anxiety: 4 items, physical problems: 2 items, trauma: 2 items); life/social functioning (close relationships: 4 items, social relationships: 4 items, general functioning: 4 items), and risk to self and others (6 items). Higher scores indicate higher levels of distress. To distinguish between clinical and non-clinical cut-off values, the four dimensions (scales for both males and females) indicated in the original validation and the Italian version (Evans et al., 2002; Palmieri et al., 2009) will be considered.
Academic motivation | before and after the psychological intervention, up to 7 weeks
  The Academic Motivation Scale (AMS) is a 20-item self-report questionnaire designed to evaluate the regulation of motivation based on the self-determination theory. Academic motivation is conceptualized according to the degree of autonomy on which the individual behavior is based, expressed through a continuum of increasing self-determination, from not self-determined (amotivation pole) to self-determined (autonomous regulation pole) behavior, from being externally motivated to becoming internally and autonomously driven to perform certain behaviors. The items are rated on a five-point Likert scale (0 = does not correspond at all to 7 = corresponds exactly) and distributed in five subscales--amotivation, external regulation, introjected regulation, identified regulation, and intrinsic motivation. Scores frange from 0 to 140. High score subscale indicates higher endorsement of that motivation type.

SECONDARY OUTCOMES:
Emotion regulation ability | before and after the treatment, up to 7 weeks
  The Difficulty in Emotion Regulation Scale (DERS) is a 36-item multi-dimensional self-report measure of emotion dysregulation and emotion self-regulation strategies. The total scores range from 36 to 180, with higher scores indicating more difficulty in the emotion regulation component measured
perceived loneliness | before and after the intervention, up to 7 weeks
  The University of California-Los Angeles (UCLA) Loneliness Scale version 3 (LS3) is a 20-item self-report measure of an individual's subjective feelings of loneliness. Higher scores indicate greater loneliness. A total score ≥ 47 will be considered indicative of higher-than-normal levels of loneliness.
drop-out intention | before and after the intervention, up to 7 weeks
  Students' intentions to continue or to drop out of the academic course will be measured with self-reported questions. For the present study, the Italian version, which consists of 4 items asking students how often they have thought about not continuing their university degree courses, will be adopted. Scores frange from 4 to 20. Higher scores indicate a greater intention to drop out.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania, Caserta, Italy

IPD SHARING:
Plan to Share IPD: Undecided
only, if requested

REFERENCES:
- [Background] Beiter R, Nash R, McCrady M, Rhoades D, Linscomb M, Clarahan M, Sammut S. The prevalence and correlates of depression, anxiety, and stress in a sample of college students. J Affect Disord. 2015 Mar 1;173:90-6. doi: 10.1016/j.jad.2014.10.054. Epub 2014 Nov 8. PMID 25462401
- [Background] Batra K, Sharma M, Batra R, Singh TP, Schvaneveldt N. Assessing the Psychological Impact of COVID-19 among College Students: An Evidence of 15 Countries. Healthcare (Basel). 2021 Feb 17;9(2):222. doi: 10.3390/healthcare9020222. PMID 33671363
- [Background] Auerbach RP, Alonso J, Axinn WG, Cuijpers P, Ebert DD, Green JG, Hwang I, Kessler RC, Liu H, Mortier P, Nock MK, Pinder-Amaker S, Sampson NA, Aguilar-Gaxiola S, Al-Hamzawi A, Andrade LH, Benjet C, Caldas-de-Almeida JM, Demyttenaere K, Florescu S, de Girolamo G, Gureje O, Haro JM, Karam EG, Kiejna A, Kovess-Masfety V, Lee S, McGrath JJ, O'Neill S, Pennell BE, Scott K, Ten Have M, Torres Y, Zaslavsky AM, Zarkov Z, Bruffaerts R. Mental disorders among college students in the World Health Organization World Mental Health Surveys. Psychol Med. 2016 Oct;46(14):2955-2970. doi: 10.1017/S0033291716001665. Epub 2016 Aug 3. PMID 27484622
- Available data/document: Informed Consent Form — https://docs.google.com/forms/d/e/1FAIpQLScX9N2R8xP62390ly7vV8Ixyy_yfQsUUmUG3QCm_M-ZriXAnA/viewform